CLINICAL TRIAL: NCT04045834
Title: Study of the Diagnostic Value of Hybrid PET/MR and PET/CT in Neuroendocrine Diseases and Tumor Induced Osteomalacia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xiaoli Lan, Director of the Department of nuclear medicine, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Other Study IDs: XLan-S1002
Record Dates: First submitted 2019-08-04; First posted 2019-08-06 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: PET / CT; PET / MR; Neuroendocrine Tumors; Osteomalacia
MeSH Terms: conditions — Neuroendocrine Tumors; Osteomalacia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: 68Ga-DOTA-TATE PET/MR and PET/CT imaging — Intravenous access is established in advance, intravenous bolus injection, 68Ga-DOTA-TATE dose is about 2 MBq/kg body weight (0.054 mCi/kg) up to 200 MBq (5.4 mCi), 18F-FDG dose is about 3.7-5.4 MBq/kg (0.1 -0.15 mCi/kg), rinsed with 0.9% saline, and hydrated after drinking more water.

SUMMARY:
Neuroendocrine tumors (NETs) are rare neoplasms arising from the diffuse endocrine system and spreading throughout the different organs and tissues of the body. Tumor-induced osteomalacia (TIO) , is a rare, serious paraneoplastic syndrome primarily derived from a benign tumor of mesenchymal tissue. NETs and mesenchymal tumors are often insidious and are undetectable by conventional imaging techniques including ultrasound, computed tomography and magnetic resonance, while a permanent cure will rely on exact localization and completely removal of the tumor.

Positron emission tomography (PET) provides a valuable tool for the diagnosis and differential diagnosis, staging, efficacy evaluation and recurrence monitoring of various tumors. NETs and mesenchymal tumors overexpress somatostatin receptors (SSTRs), so molecular imaging using radiolabeled somatostatin analogues may be one of the best ways to detect the occult tumors. Recently, somatostatin analogue labelled with gallium-68 (68Ga-DOTA-TATE) as a novel positron tracer has shown to be effective for the detection of NETs and mesenchymal tumors. In this prospective study, the investigators will use the most advanced imaging equipment, integrated PET/MR，and PET / CT with specific imaging agent 68Ga-DOTA-TATE and conventional imaging agent [F-18]fluorodeoxyglucose to image patients suspected or confirmed NETs and TIO, the aim is to explore the value of hybrid PET/MR and PET/CT in neuroendocrine diseases and TIO.

DETAILED DESCRIPTION:
Neuroendocrine tumors (NETs) are rare neoplasms arising from the diffuse endocrine system and spreading throughout the different organs and tissues of the body. Tumor-induced osteomalacia (TIO), is a rare, serious paraneoplastic syndrome primarily derived from a benign tumor of mesenchymal tissue. NETs and mesenchymal tumors are often insidious and are undetectable by conventional imaging techniques including ultrasound, computed tomography and magnetic resonance, while a permanent cure will rely on exact localization and completely removal of the tumor.

Positron emission tomography (PET) provides a valuable tool for the diagnosis and differential diagnosis, staging, efficacy evaluation and recurrence monitoring of various tumors. NETs and mesenchymal tumors overexpress somatostatin receptors (SSTRs), so molecular imaging using radiolabeled somatostatin analogues may be one of the best ways to detect the occult tumors. Recently, somatostatin analogue labelled with gallium-68 (68Ga-DOTA-TATE) as a novel positron tracer has shown to be effective for the detection of NETs and mesenchymal tumors. In this prospective study, the investigators will use the most advanced imaging equipment, integrated PET/MR，and PET / CT with specific imaging agent 68Ga-DOTA-TATE and conventional imaging agent [F-18] fluorodeoxyglucose to image patients. For patients suspected of or diagnosed with NETs and TIO, the investigators aim to evaluate the roles of integrated PET/MR and PET/CT in differential diagnosis, detecting primary and metastatic lesions, guilding biopsy, staging and determining treatment plan prior to treatment; for patients with a history of NETs and TIO, the aim is to evaluate the value of integrated PET/MR and PET/CT for treatment response assessment, detection of recurrences and metastatic lesions; for patients with inoperable and metastatic NETs, the aim is to find the value of integrated PET/MR and PET/CT in assessing the expression level of SSTRs to guide peptide receptor radionuclide therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected or confirmed NETs or patients with suspected TIO

Exclusion Criteria:

* Acute systemic diseases and electrolyte disorders.
* Pregnant or lactating women.
* Participated in other clinical trials within 4 weeks before the start of the study.

Ages: 20 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: About 90% of NETs, such as pancreatic endocrine tumors, pheochromocytoma, paraganglioma, gastrointestinal carcinoid, bronchial carcinoid, medullary thyroid carcinoma, small cell lung cancer, pituitary adenoma, some non-NETs (meninga) Tumor, astrocytoma, breast cancer, etc. have high expression of somatostatin receptor (SSTR).
  TIO tumors are often derived from benign tumors of mesenchymal tissue, mostly located in bone or soft tissue, hiding in location, slow growth, and difficult to be found, making diagnosis difficult. According to reports in the literature, most of these tumors are positive for SSTR expression, and somatostatin receptor PET/CT imaging can locate lesions, which is a good method for screening TIO and has high specificity.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-05-05 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of diagnosis and staging | up to 2 years
  The presence of non-physiological uptake or uptake in a tissue structure can be considered pathological. The signal intensity of PET indicates the presence and density of SSTR in the tissue. The lesion intake is higher than the liver and is classified as clearly positive. The lesion and the surrounding normal tissue ROI, measure the SUV, and calculate the T/B ratio. Special attention should be paid to the analysis of the causes of false positives and false negative results.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoli Lan, PhD, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- China, Hubei Province, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided